CLINICAL TRIAL: NCT01445418
Title: A Phase I Study With an Expansion Cohort of the PARP Inhibitor AZD2281 (KU-0059436) Combined With Carboplatin in Breast and Ovarian Cancer in BRCA1/2 Mutation Carriers (Familial Breast and Ovarian Cancer) and Sporadic Triple Negative Breast Cancer and Ovarian Cancer
Brief Title: AZD2281 Plus Carboplatin to Treat Breast and Ovarian Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 080092; 08-C-0092; NCT00647062 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-10-22 (Actual); Status verified 2019-10-18

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Genetic; BRCA; Ovarian Cancer, sporadic epithelial ovarian cancer; Breast Cancer, triple negative breast cancer; Metastatic; Breast Cancer; Ovarian Cancer
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Triple Negative Breast Neoplasms; Neoplasm Metastasis | interventions — Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Standard dose escalation
  Interventions: Drug: AZ2281 + Carboplatin
- Arm 2 (Experimental): Expanded cohort
  Interventions: Drug: AZ2281 + Carboplatin

INTERVENTIONS:
Drug: AZ2281 + Carboplatin — Cohort 1: Dose escalation: AZD2281 po bid qd + IV carboplatin D8 of each 21-day cycle.; Cohort 2: Expanded cohort treated at the MTD of the combination identified in Cohort 1.

SUMMARY:
Background:

* Carboplatin is approved by the Food and Drug Administration to treat cancer.
* AZD2281 is an experimental drug in a class of agents called PARP inhibitors. PARP is a protein that is -involved in repairing DNA damage; PARP inhibitors interfere with that process.

Objectives:

* To determine the optimum doses of AZD2281 and carboplatin that can safely be used in patients with breast and ovarian cancer.
* To evaluate the response of the tumor to the drug combination and determine the side effects of the treatment.

Eligibility:

-Patients 18 years of age or older with breast or ovarian cancer who have a family history of cancer or who have a BRCA1 or BRCA2 mutation.

Design:

* In this dose escalation study, the first small group of patients receives the smallest study doses of AZD2281 and carboplatin. Subsequent groups receive incrementally higher doses of first AZD2281 and then carboplatin as long as the preceding group has not experienced unacceptable side effects. When the highest safe dose is determined, additional patients receive that dose.
* Patients receive treatment in 21-day cycles as follows: AZD2281 by mouth twice a day every day; carboplatin thorough a vein on day 8 of each cycle. Treatment may continue until it is no longer beneficial.
* Evaluations during treatment include the following:
* Physical examination 1 week after starting treatment and then every 3 weeks.
* Blood tests weekly for the first 4 weeks of treatment and then every 3 weeks.
* CT scans or other imaging tests such as ultrasound or MRI every 6 weeks to evaluate the tumor.

DETAILED DESCRIPTION:
Background:

AZD2281 (KU-0059436) is an oral PARP-1 and PART-2 inhibitor that affects tumor growth by impairing the ability of the cell to repair damaged DNA. Carboplatin causes covalent cross-linking of DNA with stalled replication forks that would usually be repaired through nucleotide excision repair and homologous recombination (HR).

Sporadic breast (triple negative) and ovarian cancers have been shown to exhibit a BRCA1-like phenotype.

BRCA1/2 proteins have a critical function in the homologous DNA repair pathway. BRCA1/2 mutation carriers are at high risk for breast and ovarian cancer, and increased risk of pancreatic cancer and prostate cancer. Mutation carriers have been shown to have increased susceptibility to DNA damaging agents, such as the platinums.

BRCA1/2 deficient cells have been shown to be sensitive to PARP inhibition alone and in combination with DNA damaging agents.

Combining these two agents in a background of impaired HR in BRCA1/2 mutation potitive malignancies may result in synergistic anti-tumor effect.

Objectives:

Determine the safety and toxicity of the combination of AZD2281 and carboplatin in BRCA1/2-associated or familial recurrent breast and ovarian cancer patients (cohort 1, Group A), non-high risk serous ovarian cancer patients (Group B), and non-high risk triple negative breast cancer patients (Group C).

Determine pharmacodynamics, estimates of biochemical changes in the apoptosis and PARP signal transduction pathways in tumor and stromal cells in response to treatment of an expansion cohort (cohort 2) at the MTD in a pilot fashion.

Eligibility:

Adults with breast or ovarian CA that is metastatic or unresectable and for which standard curativetherapies do not exist or are no longer effective.

Documented deleterious BRCA1/2 mutation or a BRCAPRO score of greater than or equal to 30%.

Non-high risk serous ovarian cancer (negative family history, BRCAPRO score of less than or equal to 20% or negative BRCA1/2 mutation test).

Documented ER negative, PR negative, Her2neu negative breast cancer (negative family history and/or BRCAPRO score less than or equal to 10% (or negative BRCA1/2 mutation test).

Patients must be off prior chemotherapy, radiation therapy, hormonal therapy, or biological therapy for at least 4 weeks.

All patients enrolling in cohort 2 must have at least one lesion amenable to biopsy.

ECOG performance status 0-2 and adequate organ and marrow function.

Design:

Patients will receive AZD2281 for days 1-7 of each 21 day cycle to maximize PARP inhibition with carboplatin administration on day 2. Carboplatin will then be administered q3weeks and with continuation AZD2281 BID on days 1-7 of each 21 day cycle.

AZD2281 or carboplatin will be escalated sequentially in Cohort 1 (Groups A, B, and C), and after the maximum tolerated dose is determined, Cohort 2 will be enrolled for assessment of translational endpoints.

Patients will be evaluated for toxicity in clinic every 3 weeks and every other cycle for response using RECIST criteria. The clinic visit will be changed to every 4 weeks when patients continue to stay on the study longer than two years with no or minimal disease. Imaging studies will be obtained every 3 cycles for patients who stay on the study longer than four years. The clinic visit will be changed to every two months (+/- 7 days) and the imaging studies will be obtained every four months (+/- 7 days) for patients who stay on the study longer than five years.

Tumor biopsies and plasma and serum samples will be obtained from patients in Cohort 2 before treatment (biopsy mandatory), prior to treatment on cycle 2, day 1, and at time of disease progression (biopsies optional). Tumor biopsies (optional) will also be taken from "super responders" in Cohort 1 who have had a durable response longer than two years.

A minimum of 84 and a maximum of 101 patients will be needed to achieve the objectives of the trial.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have breast and/or epithelial ovarian cancer, primary peritoneal cancer, and/or fallopian tube cancer histologically or cytologically confirmed at the NCI that is metastatic or unresectable and for which standard curative measures do not exist or are no

longer effective.

All patients in cohort 1 must have measurable and/or evaluable disease.

Patients in the expansion cohort 2 must have safely biopsible disease as determine by an interventional radiologist and must agree to the first mandatory biopsy (the other two biopsies optional).

Breast cancer patients with locally advanced, unresectable disease must have been previously treated with standard therapy.

There is no limit on number of prior therapy.

Patients must be at least 6 months from their last platinum exposure.

Platinum-resistant patients may participate.

Patients with allergic reaction to platinums (up to and including grade 3 without a reaction protocol, and up to and including grade 2 in the face of pretrement, but not graduated treatment exposure) are still eligible.

Age greater than or equal to 18 years.

ECOG performance status less than or equal to 2 (Karnofsky greater than or equal to 60%).

Life expectancy greater than 3 months.

Patients must have normal organ and marrow function as defined below:

* hemoglobin greater than or equal to 10g/dL
* leukocytesgreater than or equal to 3,000/mcL
* absolute neutrophil count greater than or equal to 1,500/mcL
* platelets greater than or equal to 100,000/mcL
* total bilirubin less than or equal to upper limit of normal (ULN) in the absence of Gilbert s syndrome
* AST(SGOT)/ALT(SGPT) less than or equal to 2.5 X ULN
* creatinine clearance greater than or equal to 60 mL/min by 24-hour urine

OR

* serum creatinine less than or equal to 1.5 mg/dl
* corrected or Ionized Calcium less than or equal to ULN
* potassium within normal limits

A documented deleterious BRCA 1/2 germline mutation or BRCAPRO score of greater than or equal to 30% for patients enrolling in Group A.

For patients enrolling in the sporadic serous epithelial ovarian cancer group, Group B, a negative family history (BRCAPRO score less than or equal to 20% or negative BRCA1/2 mutation test).

For patients enrolling in the triple negative breast cancer (ER-/PR- /Her2-) group, Group B, a negative family history and /or BRCAPRO score less than or equal to 10% or negative BRCA1/2 mutation test).

The effects of AZD on the developing human fetus are unknown. For this reason and because platinum agents are known to be teratogenic, men and women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately, Patients of child-bearing potential should continue on contraception for at least three months following the last dose of therapy on study.

Toxicities from previous cancer therapies must have recovered to grade 1 (defined by CTC 3.0). Chronic stable grade 2 peripheral neuropathy secondary to neurotoxicity from prior therapies may be considered on a case by case basis by the Principal Investigator. No patients with functional impairment due to neuropathy will be eligible for the study. Hypomagnesemia will not be considered an exclusion criteria. Magnesium levels will be monitored and replaced as clinically indicated. Ability to understand and the willingness to sign a written informed consent document.

Female patients with reproductive potential must have a negative urine or serum pregnancy test within 4 days prior to the start of the study.

EXCLUSION CRITERIA:

Patients who have had chemotherapy, biological therapy, hormonal therapy (with the exception of raloxifene or others approved for bone health) or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study.

Patients may not be receiving any other investigational agents or had them in the previous 28 days.

Patients with known brain metastases diagnosed within 1 year should be excluded from this clinical trail because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurologic and other adverse events.

---Patients with brain metastases diagnosed greater than 1 year prior to study entry are eligible if they received sterilizing therapy to the CNS (resection or radiation) and have been CNS recurrence-free for a full 1-year period.

Clinically significant bleeding.

Inability to swallow pills.

Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Pregnant and breast-feeding women.

HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with AZD2281. In addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy such as carboplatin.

Previous treatment with PARP inhibitor.

Major surgery within the past 28 days.

Patients with locally advanced breast tumors presenting for their initial therapy, or patients with local (only in breast or chest wall) recurrence only will not be eligible for this trial

For subjects in the dose-expansion cohorts, history of prior invasive malignancies within the past 5 years (with the exception of non-melanomatous skin cancers, non-invasive bladder cancer, stage I endometrial cancer or cervical cancer cured by surgical resection).

Patients with a history of grade 4 allergic reaction to platinums

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2008-05-12; Primary Completion 2014-09-02 (Actual); Study Completion 2019-10-18 (Actual)

PRIMARY OUTCOMES:
Safety/Toxicity | End of treatment
  Determine the safety and toxicity of the combination of AZD2281 (KU- 0059436) and carboplatin in recurrent BRCA1/2-associated or familial breast and ovarian cancer patients, in recurrent low genetic risk serous ovarian cancer patients, and in recurrent low genetic risk triple negative breast cancer patients.

SECONDARY OUTCOMES:
Assess clinical activity of the combination; Determine biochemical changes in the poly(ADP-ribose) polymerase (PARP) and H2AX activity in mononuclear cells and in tumor in response to treatment | End of treatment
  Assess clinical activity of the combination; Determine biochemical changes in the poly(ADP-ribose) polymerase (PARP) and H2AX activity in mononuclear cells and in tumor in response to treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jung-Min Lee, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Alderson T. New targets for cancer chemotherapy--poly(ADP-ribosylation) processing and polyisoprene metabolism. Biol Rev Camb Philos Soc. 1990 Nov;65(4):623-41. doi: 10.1111/j.1469-185x.1990.tb01240.x. No abstract available. PMID 2124932
- [Background] Audebert M, Salles B, Calsou P. Involvement of poly(ADP-ribose) polymerase-1 and XRCC1/DNA ligase III in an alternative route for DNA double-strand breaks rejoining. J Biol Chem. 2004 Dec 31;279(53):55117-26. doi: 10.1074/jbc.M404524200. Epub 2004 Oct 21. PMID 15498778
- [Background] Berger NA, Adams JW, Sikorski GW, Petzold SJ, Shearer WT. Synthesis of DNA and poly(adenosine diphosphate ribose) in normal and chronic lymphocytic leukemia lymphocytes. J Clin Invest. 1978 Jul;62(1):111-8. doi: 10.1172/JCI109094. PMID 659624
- [Derived] Shamseddine AI, Farhat FS. Platinum-based compounds for the treatment of metastatic breast cancer. Chemotherapy. 2011;57(6):468-87. doi: 10.1159/000334093. Epub 2012 Jan 10. PMID 22248721